CLINICAL TRIAL: NCT02187965
Title: Impact of Muscle Fat Accumulation on the Genomic Profile of Skeletal Muscle in Older Adults
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Purdue University
Other Study IDs: 1107011060
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2011-08

CONDITIONS: Intermuscular Adipose Tissue Quantification

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — muscle tissue, RNA

SUMMARY:
Subjects were asked to come to the Purdue facilities after an overnight fast on 2 different testing days for 2.5 hours each day. On one day the subjects participated in blood pressure and body weight measurements as well as a muscle biopsy from the thigh. On the second day the subjects underwent an MRI and MRS scan of the thigh and calf.

ELIGIBILITY:
Inclusion Criteria:

* 60-80 years old, men and women, normal body weight or obese,

Exclusion Criteria:

* Certain medical conditions could have placed them at risk

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: normal weight and obese older adults
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
MRI | 1 day
  To determine the within day reproducibility of MRI scans for intermuscular adipose tissue (IMAT) quantification in older men and women.

SECONDARY OUTCOMES:
genomic profile | 1 day
  To examine the influence of IMAT accumulation on the genomic profile of skeletal muscle of normal weight or obese adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States